CLINICAL TRIAL: NCT06014190
Title: A Phase 2 Study of HS-20089 for Injection in Patients With Recurrent or Metastatic Ovarian Cancer and Endometrial Cancer
Brief Title: HS-20089 in Patients With Ovarian Cancer and Endometrial Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-20089-201
Record Dates: First submitted 2023-08-16; First posted 2023-08-28 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer; Endometrial Cancer
Keywords: HS-20089; B7-H4; Antibody-drug Conjugate; Ovarian Cancer; Endometrial Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 at 4.8 mg/kg of HS-20089 (Phase 2a) (Experimental): Patients in cohort 1 of phase 2a will be randomly assigned to receive HS-20089 at 4.8 mg/kg or 5.8 mg/kg.
  Interventions: Drug: HS-20089
- Cohort 1 at 5.8 mg/kg of HS-20089 (Phase 2a) (Experimental): Patients in cohort 1 of phase 2a will be randomly assigned to receive HS-20089 at 4.8 mg/kg or 5.8 mg/kg.
  Interventions: Drug: HS-20089
- Cohort 2 at 5.8 mg/kg of HS-20089 (Phase 2a) (Experimental): Patients in cohort 2 of phase 2a will receive HS-20089 at 5.8 mg/kg.
  Interventions: Drug: HS-20089
- Cohort 3 at 5.8 mg/kg of HS-20089 (Phase 2a) (Experimental): Patients in cohort 3 of phase 2a will receive HS-20089 at 5.8 mg/kg.
  Interventions: Drug: HS-20089
- Cohort 4 at 5.8 mg/kg of HS-20089 (Phase 2a) (Experimental): Patients in cohort 4 of phase 2a will receive HS-20089 at 5.8 mg/kg.
  Interventions: Drug: HS-20089
- Recommended dose of HS-20089 (Phase 2b) (Experimental): Patients of phase 2b will receive HS-20089 at recommended dose.
  Interventions: Drug: HS-20089

INTERVENTIONS:
Drug: HS-20089 — All patients will receive intravenous HS-20089 once every three weeks (Q3W) until experiencing objective disease progression (except for study drug treatment beyond progression) or meeting other protocol-specified criteria of study treatment discontinuation.

SUMMARY:
HS-20089 is an investigational antibody-drug conjugate (ADC) composed of a humanized IgG1 anti-B7-H4 monoclonal antibody conjugated to the topoisomerase I inhibitor payload via a protease-cleavable linker, with an average drug-to-antibody ratio of about 6.

This is a phase 2, open-label, multi-center study to evaluate the efficacy, safety, pharmacokinetics (PK) and immunogenicity of HS-20089 as monotherapy in patients with recurrent or metastatic ovarian cancer and endometrial cancer.

DETAILED DESCRIPTION:
This is a phase 2, open-label, multi-center study composed of two parts: phase 2a and phase 2b.

Phase 2a: This part of study will be conducted in the following four cohorts: Cohort 1: Patients with platinum-resistant ovarian cancer, fallopian tube cancer or primary peritoneal cancer. Cohort 2: Patients with recurrent or metastatic endometrial cancer who have progressed on or are intolerant to at least one line of standard platinum-based chemotherapy. Cohort 3: Patients with platinum-sensitive ovarian cancer, fallopian tube cancer or primary peritoneal cancer who have progressed on or are intolerant to at least two lines of standard platinum-based chemotherapy. Cohort 4: Patients with other advanced solid tumors who have progressed on or are intolerant to established standard therapies. Patients in cohort 1 will be randomly assigned 1:1 to receive HS-20089 at 4.8 mg/kg or 5.8 mg/kg and patients in the other three cohorts will receive HS-20089 at 5.8 mg/kg.

Phase 2b: This part of study will be conducted in the following two cohorts: Cohort 1: Patients with platinum-resistant ovarian cancer, fallopian tube cancer or primary peritoneal cancer. Cohort 2: Patients with recurrent or metastatic endometrial cancer who have progressed on or are intolerant to at least one line of standard platinum-based chemotherapy. The cohorts may be adjusted based on the observed clinical results, translational medicine data and research progress in the field. All patients will receive HS-20089 at the recommended dose (RD) determined by accumulated research data.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 years or older (≥18 years).
2. Patients diagnosed with recurrent or metastatic ovarian cancer, endometrial cancer or other solid tumors.
3. Subjects have at least one target lesion as assessed per the RECIST 1.1. Patients with only brain and/or bone lesions as target lesions are ineligible.
4. Tumor tissue from a newly obtained biopsy (FFPE tumor tissue blocks or slides are acceptable) is required. If the newly obtained biopsy is not feasible, newly obtained FFPE slides cut from archival tumor tissue blocks within 2 years prior to the first dose of study drug are acceptable.
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 to 1 and no deterioration within 2 weeks before the first dose.
6. Have a life expectancy of at least 12 weeks.
7. Female subjects of childbearing potential are willing to take appropriate contraceptive measures and should not breastfeed from signing the informed consent until 6 months after the last dose; male subjects must agree to use barrier contraception (i.e. condoms) from signing the informed consent to 6 months after the last dose.
8. Female subjects must have a negative pregnancy test within 7 days prior to the first dose (for subjects with tumor related abnormal elevation of human chorionic gonadotropin [HCG], an ultrasound of uterus and appendages should be performed within 7 days prior to the first dose to rule out pregnancy), or demonstrate no risk for pregnancy.
9. Subject must be voluntarily enrolled in this clinical trial, be able to understand the study procedures and to sign written informed consent.

Exclusion Criteria:

1. Have received or is currently receiving the following treatment:

   1. B7-H4-targeted therapies.
   2. Have received any of cytotoxic chemotherapy drugs, investigational drugs, anti-tumor traditional Chinese medicines or other anti-tumor drugs (including endocrine therapy, molecular targeted therapy, biotherapy, etc.) within 14 days prior to the first dose of study drug; or need to continue these drugs during the study.
   3. Have received macromolecular antitumor drugs (including immunotherapy, such as monoclonal antibodies and bispecific antibodies) within 28 days prior to the first dose of study drug.
   4. Have received locoregional radiation therapy within 2 weeks prior to the first dose of study drug; more than 30% of bone marrow irradiation or wide-field radiation therapy within 4 weeks prior to the first dose of study treatment.
   5. Major surgery (such as craniotomy, thoracotomy or laparotomy, etc.) within 4 weeks prior to the first dose of study treatment.
   6. Use of strong inhibitors or inducers of CYP3A4, CYP2D6, P-gp, or BCRP, or sensitive substrates of CYP3A4, CYP2D6, P-gp, or BCRP with narrow therapeutic window within 7 days prior to the first dose of study drug; or in need of continuing treatment with these drugs during the study.
   7. Current use of drugs known to prolong the QT interval or potentially cause torsades de pointes; or need to continue these medications during the study.
2. Presence of Grade ≥ 2 toxicities as per Common Terminology Criteria for Adverse Events (CTCAE version 5.0) due to prior anti-tumor therapy (except alopecia and residual neurotoxicity).
3. Presence of pleural/abdominal effusion requiring clinical intervention.
4. Known history of prior malignancy.
5. Evidence of brain metastasis, unless meeting all of the following criteria:

   1. Asymptomatic; medically stable for at least four weeks prior to the first dose;
   2. No steroid treatment required for at least two weeks prior to the first dose;
   3. No stereotactic radiation therapy, whole brain radiotherapy, and/or neurosurgical resection within 4 weeks prior to the first dose;
   4. No history of intracranial or spinal hemorrhage;
   5. Have at least one target lesion other than CNS lesion according to RECIST v1.1;
6. Inadequate bone marrow reserve or hepatic/renal functions.
7. Cardiological examination abnormality.
8. Severe, uncontrolled or active cardiovascular disorders.
9. Serious or poorly controlled diabetes.
10. Serious or poorly controlled hypertension.
11. Clinically significant bleeding symptoms or significant bleeding tendency within 1 month prior to the first dose of study treatment.
12. Serious arteriovenous thromboembolic events within 3 months prior to the first dose of study treatment.
13. Serious infections within 4 weeks prior to the first dose.
14. Have received systemic glucocorticoid therapy for more than 30 days within 30 days prior to the first dose study treatment, or require chronic (≥ 30 days) use of systemic glucocorticoids during the study, or have other acquired, congenital immunodeficiency disorders, or a history of organ transplantation.
15. Presence of active infectious diseases such as hepatitis B, hepatitis C, tuberculosis, syphilis, or human immunodeficiency virus infection, etc.
16. Current hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh Class B or more severe cirrhosis.
17. Any moderate or severe lung diseases that may interfere with the detection and treatment of drug-related pulmonary toxicity or may seriously affect respiratory function.
18. History of severe neurological or psychiatric disorder.
19. Pregnant or breast-feeding women or women who intend to become pregnant during the study.
20. Attenuated live vaccination within 4 weeks prior to the first dose.
21. Allergies or hypersensitivity reactions within 4 weeks prior to the first dose. History of severe allergies (e.g., anaphylactic shock), or severe infusion-related reactions. Allergy or hypersensitivity to any component of HS-20089.
22. Subjects unlikely to comply with study procedures, restrictions and requirement as determined by the investigator.
23. Subjects with any condition that jeopardizes the safety of the patient or interferes with the assessment of the study, as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) assessed by investigators according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | From the first dose up to disease progression or withdrawal from study, whichever came first, assessed up to 24 months.
  ORR is defined as the percentage of participants who achieved a best overall response (BOR) of confirmed complete response (CR) or partial response (PR), assessed by investigators based on RECIST 1.1.

SECONDARY OUTCOMES:
ORR assessed by independent review committee (IRC) according to RECIST 1.1 | From the first dose to disease progression or withdrawal from study, whichever came first, assessed up to 24 months.
  ORR is defined as the percentage of participants who achieved a BOR of confirmed CR or PR, assessed by IRC based on RECIST 1.1.
Duration of response (DoR) assessed by investigators and IRC according to RECIST 1.1 | From the first dose to disease progression or withdrawal from study, whichever came first, assessed up to 24 months.
  DoR is defined as the period from the first occurrence of CR or PR to progressive disease (PD) or death of any cause. If no PD or death after CR/PR, the cut-off date of progression-free survival (PFS) will be used.
Disease control rate (DCR) assessed by investigators and IRC according to RECIST 1.1 | From the first dose to disease progression or withdrawal from study, whichever came first, assessed up to 24 months.
  DCR is defined as the percentage of participants with BOR of confirmed CR, PR and stable disease (SD).
Progression-free survival (PFS) assessed by investigators and IRC according to RECIST 1.1 | From the first dose or randomization to disease progression or withdrawal from study, whichever came first, assessed up to 24 months.
  PFS is defined as the time from first dose or randomization (if any) to PD or death of any cause.
Overall survival (OS) | From the first dose or randomization to death or withdrawal from study, whichever came first, assessed up to 24 months.
  OS is defined as the time from the first dose or randomization (if any) to death of any cause.
ORR assessed by investigators (combined criteria incorporating RECIST 1.1 and Gynecological Cancer Intergroup [GCIG]) CA-125 criteria; Ovarian cancer only) | From the first dose to disease progression or withdrawal from study, whichever came first, assessed up to 24 months.
  Defined as the proportion of subjects with confirmed CR or PR before progression as assessed by incorporating both RECIST 1.1 and GCIG CA-125 criteria.
CA-125 response rate assessed by investigators according to GCIG CA-125 criteria (ovarian cancer only) | From the first dose to disease progression or withdrawal from study, whichever came first, assessed up to 24 months.
  CA-125 response rate is defined as the proportion of subjects with GCIG CA-125 criteria defined CA-125 response, which will be assessed in a subset of subjects with a baseline CA-125 level of at least twice the ULN as evaluable.
Incidence and severity of adverse events (AEs) | From the first dose to 90 days after the end of treatment.
  AEs will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0. The incidence and severity of AEs will be calculated and summarized.
Observed maximum plasma concentration (Cmax) of HS-20089 | From pre-dose to 14 days after the first dose of HS-20089 on Cycle 1 (each cycle is 21 days).
  Cmax will be obtained following administration of the first dose of HS-20089 during the first cycle.
Time to reach maximum plasma concentration (Tmax) of HS-20089 following the first dose | From pre-dose to 14 days after the first dose on Cycle 1 (each cycle is 21 days).
  Tmax will be obtained following administration of the first dose of HS-20089 during the first cycle.
Area under plasma concentration versus time curve from zero to last sampling time (AUC0-t) following the first dose of HS-20089 | From pre-dose to 14 days after the first dose on Cycle 1 (each cycle is 21 days).
  Area under the plasma concentration versus time curve from time zero to the last sampling time when the concentration is no less than the lower limit of quantification (LLQ). AUC0-t will be calculated according to the mixed log-linear trapezoidal rule.
Area under the plasma concentration versus time curve from time zero to infinity (AUC0-∞) after single dose of HS-20089 | From pre-dose to 14 days after the first dose on Cycle 1 (each cycle is 21 days).
  AUC0-∞ will be calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast/ λz, where Clast is the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the LLQ and λz is the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Percentage of participants with antibodies to HS-20089 in serum | From the first dose to 90 days after the end of treatment.
  Serum samples will be collected for the determination of anti-drug antibody (ADA) at designated time points.

CONTACTS AND LOCATIONS:
Overall Officials: Lingying Wu, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (28):
- China (28):
  - Anhui Provincial Cancer Hospital, Hefei, Anfei
  - Lingying Wu, Beijing, Beijing Municipality
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing University cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-Sen Memorial Hospital Sun Yat-Sen University, Guangzhou, Guangdong
  - Guangxi Cancer Hospital, Nanning, Guangxi
  - Hainan General Hospital, Haikou, Hainan
  - The fourth Hospital of Heibei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer University, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hosipital, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - The first Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Tianjin Medical University cancer institute & Hospital, Tianjin, Tianjin Municipality
  - Affiliated Cancer Hospital of Xinjiang Medical University, Xinjiang, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hanzhou, Zhejiang